CLINICAL TRIAL: NCT06811636
Title: Clinical and Radiographic Evaluation of Lesion Sterilization With Triple Antibiotic Paste Versus Root Canal Treatment With Calcium Hydroxide-iodoform Paste in Mandibular Primary Molars Diagnosed With Necrotic Pulp or Irreversible Pulpitis
Brief Title: Lesion Sterilization Tissue Repair and Conventional Pulpectomy in Primary Molars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Sümeyye ŞENOL, Research Assistant, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CanakkaleOMU1
Record Dates: First submitted 2025-01-09; First posted 2025-02-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-08

CONDITIONS: Pulpitis - Irreversible; Pulp Necroses; Root Canal Infection
Keywords: Lesion Sterilization Tissue Repair; Conventional Pulpectomy
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Lesion sterilization and tissue repair
  Interventions: Procedure: Lesion sterilization and tissue repair
- control group (Active Comparator): Conventional pulpectomy
  Interventions: Procedure: Conventional pulpectomy

INTERVENTIONS:
Procedure: Lesion sterilization and tissue repair — Lesion sterilization and tissue repair therapy performed with a triple antibiotic mixture.
  Arms: study group
Procedure: Conventional pulpectomy — Conventional pulpectomy with calcium hydroxide-iodoform based root canal paste.
  Arms: control group

SUMMARY:
The aim of this study was to compare the clinical and radiographic success of conventional root canal treatment and lesion sterilisation tissue repair methods in deciduous molars with necrotic or irreversible pulpitis.

DETAILED DESCRIPTION:
The study will be conducted on children aged 3-8 years who present to the Department of Pediatric Dentistry at Çanakkale Onsekiz Mart University, Faculty of Dentistry. The aim of the study is to compare the clinical and radiographic success of conventional root canal treatment using a calcium hydroxide-iodoform-based root canal paste and lesion sterilization tissue repair (LSTR) therapy using a triple antibiotic mixture of metronidazole, ciprofloxacin, and clindamycin in mandibular primary molars diagnosed with necrotic or irreversible pulpitis, meeting the inclusion and exclusion criteria.

The null hypothesis of the study is that there will be no significant difference in clinical and radiographic success between conventional root canal treatment and lesion sterilization tissue repair at any follow-up period.

The study plans to enroll 37 (thirty-seven) participants in the research group and 37 (thirty-seven) participants in the comparison group. The sample size was calculated based on the parameters derived from the study by Moura et al., which compared the clinical and radiographic success of conventional root canal treatment using zinc oxide eugenol and lesion sterilization tissue repair using a triple antibiotic paste. With a power level of 0.8, an alpha error probability of 0.05, and an effect size of 0.4020915, the required sample size was determined using the G*Power 3.0.10 software (v.3.1.9.7, Universitat Kiel, Kiel, Germany).

In the comparison group, conventional pulpectomy (root canal treatment) using a calcium hydroxide-iodoform-based root canal filling paste will be performed on the teeth. In the research group, lesion sterilization tissue repair therapy will be carried out using a triple antibiotic mixture of metronidazole, ciprofloxacin, and clindamycin.

The common procedural steps for both groups will include:

Initial clinical examination and radiographic imaging, Administration of mandibular alveolar nerve block anesthesia using lidocaine hydrochloride with a vasoconstrictor, Rubber dam isolation to minimize bacterial contamination and protect soft and hard tissues, Removal of carious enamel and cavity preparation using a sterile diamond fissure and round burs with a water-cooled handpiece, Complete removal of carious dentin and the roof of the pulp chamber using low-speed tungsten carbide round burs and diamond fissure burs, Removal of coronal pulp tissue with a sharp sterile excavator, followed by irrigation of the pulp chamber with sterile saline to remove any pulp remnants.

Following these steps, the treatment will proceed according to the assigned group as outlined below:

Research Group:

For the lesion sterilization tissue repair method, a triple antibiotic paste will be placed in the pulp chamber. In previous studies, minocycline was used in the triple antibiotic paste; however, concerns about tooth discoloration associated with tetracycline derivatives have been reported. Although minocycline and clindamycin demonstrate similar success rates, a recent systematic review highlighted that mixtures containing tetracyclines are statistically less effective than those without tetracyclines. Consequently, the American Academy of Pediatric Dentistry recommends excluding tetracyclines in antibiotic mixtures used for non-vital pulp therapy in primary teeth. Based on this recommendation, the triple antibiotic paste will be prepared using commercially available metronidazole, ciprofloxacin, and clindamycin.

The tablets' enteric coatings and capsules will be removed, and each drug will be ground into a fine powder using a mortar and pestle. The powders will be stored separately in tightly sealed containers to prevent exposure to light and moisture. Equal parts of each powder will be measured using a precision balance with five decimal places and mixed on a glass slab to achieve a 1:1:1 ratio. A liquid mixture of propylene glycol and macrogol will be prepared in equal proportions and combined with the powders to form the paste. The final consistency of the triple antibiotic paste will be adjusted to a 7:1 powder-to-liquid ratio (70% hardness).

The canal orifices will be widened by 1-2 mm using a small, low-speed round bur, and the walls of the pulp chamber will be chemically cleaned with phosphoric acid for one minute. After rinsing with sterile saline and drying with cotton pellets, the triple antibiotic paste will be applied directly to the canal orifices and the pulp chamber floor. The teeth will then be sealed with glass ionomer cement and restored with stainless steel crowns.

Comparison Group:

The root length of the teeth will be determined using diagnostic radiographs. The canals will be enlarged by 2-3 file sizes beyond the initial file size using K-type endodontic files. During canal preparation, each file will be followed by irrigation with 2 mL of 2.5% sodium hypochlorite (NaOCl). After canal preparation, the canals will be irrigated with 2.5% NaOCl and finally with saline before drying with paper points. The canals will then be filled with a calcium hydroxide-iodoform paste. The pulp chamber will be sealed with glass ionomer cement, and the teeth will be restored with stainless steel crowns.

Postoperative periapical radiographs of the treated teeth will be obtained. Clinical evaluations will be performed at 1, 3, 6, 9, 12, 18, 24, 30 and 36 months to assess clinical success, while radiographic evaluations will be conducted at 3, 6, 12, 18, 24, 30 and 36 months to assess radiographic success rates in both groups.

ELIGIBILITY:
Inclusion Criteria:

* The participant is between the ages of 3 and 8 years.
* The participant and their parent(s) have signed informed consent forms agreeing to participate in the study.
* The patient is systemically healthy.
* The patient's cooperation level is sufficient for performing the procedures.
* No history of allergic reactions to the materials and substances to be used.
* Mandibular primary molars diagnosed with pulp necrosis or irreversible pulpitis.
* Presence of endodontic-origin gingival abscess or fistula in the involved teeth.
* History of spontaneous pain.
* Presence of radiolucency in the furcation or periapical region, not exceeding one-third of the affected area.
* Presence of deep dentin caries causing pulp exposure.
* Presence of mobility at level 0 or 1 according to Miller's classification (non-pathologic).
* The tooth meets the criteria for restorability.
* Root resorption does not exceed more than four-fifths of the root.
* The tooth meets the criteria for isolation.

Exclusion Criteria:

* The participant is not between the ages of 3 and 8 years.
* The participant and/or their parent(s) have not agreed to participate in the study or have not signed the informed consent forms.
* The patient has a systemic disease.
* The patient's cooperation level is insufficient to perform the procedures.
* The patient has a history of allergic reactions to the materials and substances to be used.
* Teeth with external or internal root resorption.
* Mechanical or carious perforation of the pulp floor in the affected teeth.
* Radiolucency and bone destruction in the furcation or periapical region exceeding one-third of the affected area.
* Presence of caries that does not cause pulp exposure.
* Pathological mobility according to Miller's classification (>1 score).
* The tooth does not meet the criteria for restorability.
* Root resorption exceeds more than four-fifths of the root.
* The tooth does not meet the criteria for isolation.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical success | Follow up will be for three year with recall visits at 1, 3, 6, 12, 18, 24, 30 and 36 months.
  * Absence of spontaneous pain.
  * Absence of sensitivity to percussion using dental mirror, pain on biting.
  * Absence of swelling.
  * Absence of fistula / Exudate.
  * Absence of non-physiological mobility
Miller Classification - Tooth Mobility | 1, 3, 6, 12, 18, 24, 30, and 36 months.
  Class 0 Normal (physiologic) movement when force is applied.
  Class I Mobility greater than physiologic.
  Class II Tooth can be moved up to 1mm or more in a lateral direction (buccolingual or mesiodistal).
  Inability to depress the tooth in a vertical direction (apicocoronal).
  Class III Tooth can be moved 1mm or more in a lateral direction (buccolingual or mesiodistal).
  Ability to depress the tooth in a vertical direction (apicocoronal).
Radiographic success | Follow up will be for three year with recall visits at 1, 3, 6, 12, 18, 24, 30 and 36 months.
  * Absence of furcation or periapical radiolucency.
  * Absence of change in the extent of internal or external root resorption other than physiologic resorption.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye Şenol, R.A., Principal Investigator — Çanakkale Onsekiz Mart University; Berkant Sezer, Assoc. Prof., Principal Investigator — Çanakkale Onsekiz Mart University
Locations (1):
- Canakkale Onsekiz Mart University, Çanakkale, Kepez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In this study, we are committed to sharing our findings while ensuring the privacy and confidentiality of our participants. Therefore, we will only be disseminating aggregated statistical results derived from the data, rather than individual participant data.